CLINICAL TRIAL: NCT04413331
Title: Cohort Study of Vasculitis Patients: Longitudinal Study for the Assessment of Presentation, Comorbidities, Management, Outcomes and Damage
Brief Title: Prospective Longitudinal Cohort Study of Vasculitis Patients
Acronym: VASCO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200109
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Vasculitis
Keywords: Prospective vasculitis cohort
MeSH Terms: conditions — Vasculitis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, Peripheral blood mononuclear cells, DNA, RNA, urin, stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vasculitis: Those with systemic vasculitis
  Interventions: Other: Data collection; Other: Biological samples and data collection
- EGPA vasculitis
  Interventions: Other: Data collection; Other: Biological samples and data collection

INTERVENTIONS:
Other: Data collection — Medical data collection at M0, M3, M6, M9 and M12 then every 6 months until M60 and at each vascularitis relapse
Other: Biological samples and data collection — Biological samples at M0, M6, M12, M24 and at each relapse until M60

SUMMARY:
VASCO is a prospective observational cohort study which aim to describe the presentation, comorbidities, management, outcomes and damage of vasculitis patients, from the analysis of the clinical, biological and immunological data.

DETAILED DESCRIPTION:
Vasculitis is a group of disorders characterized by the inflammation of blood vessels, leading to an alteration of the vascular wall. The classification of vasculitides has evolved considerably over the last few decades.

In 1990, the American College of Rheumatology established a classification of the main systemic vasculitides based on clinical, biological and histological criteria. In 1994, the Chapel Hill nomenclature has been established as the reference classification system of vasculitides and vasculitides were classified according to the size of the affected vessels. The Chapel Hill nomenclature was revised in 2012, thus enabling to integrate new vasculitides and diagnostic tools.

It is proposed here to conduct a non-interventional cohort study of the different forms of vasculitis, as defined in the Chapel Hill nomenclature. By collecting data from a large number of patients followed prospectively, our objective is to describe the clinical patterns of these diseases, the presentation, management, comorbidities and outcomes, and to evaluate their possible association with some immunological, genetic and molecular parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age over 18 years),
* Patients with vasculitis, as defined in the Chapel Hill International Nomenclature as revised in 2012,
* Patients included at an active phase of the disease, either the initial flare or a relapse,
* Patients who have been informed and have signed the consent
* Pregnant and breastfeeding women may be included in the study,
* Affiliated to a social security system (beneficiary or entitled person).

Exclusion Criteria:

* Refusal of consent or inability to obtain consent,
* A patient who is insane or not entitled, for psychiatric reasons or intellectual impairment, to receive information about the protocol and to give informed consent,
* Patient under guardianship / curators
* Patient on state medical assistance (AME)
* Hemoglobin less than 7 g/dl at the time of sampling,
* Hemoglobin level less than 9 g/dl at the time of sampling if the patient has respiratory or cardiovascular disease,
* Patient weighs less than 18 kg.
* Parallel participation in an interventional protocol is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The VASCO study population includes adult patients (no age upper-limit) with vasculitis as defined in the 2012 revised Chapel Hill International Nomenclature, at an active phase of the disease, either the initial flare or a relapse. Patients will be informed by the study investigator during a visit as part of their medical follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Creation of a prospective cohort of vasculitis | 5 years
  Vasco cohort : To create of a large prospective cohort of vasculitis patients to describe the presentation, therapeutic management, comorbidities and outcomes, based on the analysis of clinical, biological and immunological data
Creation of a prospective cohort of EGPA-vasculitis | 5 years
  EGPA -Vasco cohort : To create of a large prospective cohort of vasculitis patients to describe the presentation, therapeutic management and his efficacity, comorbidities and outcomes of EGPA, based on the analysis of clinical, biological and immunological data.
  The evaluation of the response to the treatment will be based, for all the different treatments, on the ability or not to reach a prednisone dose of 4.0 mg or less, at any time (binary criterion)).
  The treatments will be used at the discretion of the referring physician in charge of the pathology, according to what is recommended in the National Diagnostic and Care Protocol (PNDS) in force.

SECONDARY OUTCOMES:
Identification of patterns of vasculitis | 5 years
  To identify possible relationships between clinical patterns of vasculitis and response to treatment, risk of glucocorticoids dependence, survival, etc.
Identification of comorbidities | 5 years
  To identify comorbidities and the impact on therapeutic management and patient outcomes
Identification of predictive and prognostic factors | 5 years
  To identify radiological, histological, pharmacological, genetic, molecular and immunological predictive and prognostic markers.
Evaluation of results reported by patients | 5 years
  Evaluate the results reported by patients (Patient Reported Outcomes, PROs) within the framework of the Community of Patients for Research (COMPARE)
Monitoring of the results reported by patients | 5 years
  Monitor the results reported by patients (Patient Reported Outcomes, PROs) within the framework of the Community of Patients for Research (COMPARE)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de médecine interne, Hôpital Cochin, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Undecided

REFERENCES:
- [Background] Leavitt RY, Fauci AS, Bloch DA, Michel BA, Hunder GG, Arend WP, Calabrese LH, Fries JF, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Wegener's granulomatosis. Arthritis Rheum. 1990 Aug;33(8):1101-7. doi: 10.1002/art.1780330807. PMID 2202308
- [Background] Lightfoot RW Jr, Michel BA, Bloch DA, Hunder GG, Zvaifler NJ, McShane DJ, Arend WP, Calabrese LH, Leavitt RY, Lie JT, et al. The American College of Rheumatology 1990 criteria for the classification of polyarteritis nodosa. Arthritis Rheum. 1990 Aug;33(8):1088-93. doi: 10.1002/art.1780330805. PMID 1975174
- [Background] Masi AT, Hunder GG, Lie JT, Michel BA, Bloch DA, Arend WP, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, et al. The American College of Rheumatology 1990 criteria for the classification of Churg-Strauss syndrome (allergic granulomatosis and angiitis). Arthritis Rheum. 1990 Aug;33(8):1094-100. doi: 10.1002/art.1780330806. PMID 2202307
- [Background] Jennette JC, Falk RJ, Andrassy K, Bacon PA, Churg J, Gross WL, Hagen EC, Hoffman GS, Hunder GG, Kallenberg CG, et al. Nomenclature of systemic vasculitides. Proposal of an international consensus conference. Arthritis Rheum. 1994 Feb;37(2):187-92. doi: 10.1002/art.1780370206. PMID 8129773
- [Background] Jennette JC, Falk RJ, Bacon PA, Basu N, Cid MC, Ferrario F, Flores-Suarez LF, Gross WL, Guillevin L, Hagen EC, Hoffman GS, Jayne DR, Kallenberg CG, Lamprecht P, Langford CA, Luqmani RA, Mahr AD, Matteson EL, Merkel PA, Ozen S, Pusey CD, Rasmussen N, Rees AJ, Scott DG, Specks U, Stone JH, Takahashi K, Watts RA. 2012 revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides. Arthritis Rheum. 2013 Jan;65(1):1-11. doi: 10.1002/art.37715. No abstract available. PMID 23045170
- [Background] van der Woude FJ, Rasmussen N, Lobatto S, Wiik A, Permin H, van Es LA, van der Giessen M, van der Hem GK, The TH. Autoantibodies against neutrophils and monocytes: tool for diagnosis and marker of disease activity in Wegener's granulomatosis. Lancet. 1985 Feb 23;1(8426):425-9. doi: 10.1016/s0140-6736(85)91147-x. PMID 2857806
- [Background] Sable-Fourtassou R, Cohen P, Mahr A, Pagnoux C, Mouthon L, Jayne D, Blockmans D, Cordier JF, Delaval P, Puechal X, Lauque D, Viallard JF, Zoulim A, Guillevin L; French Vasculitis Study Group. Antineutrophil cytoplasmic antibodies and the Churg-Strauss syndrome. Ann Intern Med. 2005 Nov 1;143(9):632-8. doi: 10.7326/0003-4819-143-9-200511010-00006. PMID 16263885
- [Background] Bligny D, Mahr A, Toumelin PL, Mouthon L, Guillevin L. Predicting mortality in systemic Wegener's granulomatosis: a survival analysis based on 93 patients. Arthritis Rheum. 2004 Feb 15;51(1):83-91. doi: 10.1002/art.20082. PMID 14872460
- See also: Related Info — https://www.vascularites.org/